CLINICAL TRIAL: NCT00362453
Title: Tai Chi Mind-Body Therapy for Knee Osteoarthritis: a Pilot Single-blind Randomized Controlled Trial
Brief Title: Tai Chi Mind-Body Therapy for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002161 (NIH); R21AT002161 (NIH)
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): The Tai Chi program was based on the classical Yang Style. Patients participated in 60-minute Tai Chi sessions twice a week for 12 weeks. Each session included warm up and review of Tai Chi principles and techniques; Tai Chi exercises; breathing techniques; and various relaxation methods. The classes were taught by a Tai Chi master with over 20 years' experience conducting Tai Chi Mind-Body exercise programs. Several modifications were developed to achieve the physical and mental goals of the study for knee OA, accommodate knee OA symptoms and limit dropouts. Subjects were instructed to practice Tai Chi at least 20 minutes a day at home and encouraged to maintain their usual physical activities, but not to participate in additional new strength training other than their Tai Chi exercises.
  Interventions: Behavioral: Tai Chi versus Attention Control
- Wellness Education and Stretching (Placebo Comparator): The wellness education and stretching program provided an active control for the attention being paid to the Tai Chi group. The control group attended two 60-minute class sessions per week for 12 weeks. Each session started with 40 minutes of didactic lessons on OA knowledge, nutrition, and physical and mental health education. The final 20 minutes consisted of stretching exercises involving the upper body, trunk and lower body, each stretch being held for 10 to 15 seconds. Participants were also instructed to practice at least 20 minutes of stretching exercises per day at home. They were encouraged to maintain their usual physical activities, but not to participate in additional strength and mind-body exercise programs other than their stretching exercise.
  Interventions: Behavioral: Tai Chi versus Attention Control

INTERVENTIONS:
Behavioral: Tai Chi versus Attention Control — 60 minutes, twice a week for 12 weeks.
  Other Names: Yang style Tai Chi

SUMMARY:
The purpose of this study was to compare the safety and effectiveness of Tai Chi with an Attention Control intervention consisting of a stretching and wellness education program involving 40 patients with osteoarthritis (OA) of the knee. We hypothesized that the participants receiving Tai Chi would show greater improvement in knee pain, physical and psychological functioning, and health-related quality of life than participants in the Attention Control group, and that the benefit would be mediated by effects on muscle function, musculoskeletal flexibility and mental health.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis in the United States, affecting 21 million older people. Symptomatic knee OA in the elderly is one of the most frequent causes of loss of independence and physical disability. There are currently no satisfactory pharmacological or non-pharmacological therapies for knee OA. New strategies to improve functional capacity, quality of life and reduce long-term disability in people with knee OA are urgently needed. Our long-term goal is to demonstrate the physical and psychological benefits of Tai Chi exercise as a complementary treatment for people with knee OA. Tai Chi is a traditional Chinese discipline with both physical and mental components that appear to benefit a variety of conditions. The physical component provides exercise that is consistent with recommendations for OA (range of motion, flexibility, muscle conditioning and aerobic cardiovascular exercise), while the mental component has the potential to increase psychological well-being, life satisfaction, and perceptions of health. These effects are especially pertinent for the treatment of older adults with knee OA.

Over a three-year period, 40 patients with symptomatic knee OA were randomly assigned to receive a 12-week Tai Chi program or stretching and wellness education program. Outcome measurements were obtained at baseline and on completion of the 12-week program, as well as 24 and 48 week follow-up periods. We compared changes in knee pain, stiffness, and physical function using the well-validated Western Ontario and McMaster Index (WOMAC), as well as clinical knee examination, lower extremity function, knee joint proprioception, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* Body Mass Index (BMI) <= 40 kg/m
* Pain on more than half the days of the past month during at least one of the following activities (walking, going up or down stairs, standing upright, or in bed at night
* Radiographic evidence of knee OA, defined as the presence of osteophytes in the tibiofemoral compartment and/or the patellofemoral compartment, as assessed on standing anterior/posterior and lateral views
* WOMAC pain subscale score, at least 1 of 5 (range 0 to 100 each) >= 40 (visual analog version)
* Physically able to participate in both the Tai Chi and stretching and education programs
* Willing to complete the 12-week study, including twice a week Tai Chi or stretching and education sessions
* Willing to abstain from Tai Chi until completion of the program, if randomized to the stretching and education sessions
* Willing to abstain from stretching and education sessions until completion of the program, if randomized to Tai Chi

Exclusion Criteria:

* Prior experience with Tai Chi or other similar types of Complementary and Alternative Medicine such as Qi gong, yoga, and acupuncture since these share some of the principles of Tai Chi
* Dementia, neurological disease, cardiovascular disease, pulmonary disease, metabolic disease, renal disease, liver disease, or other serious medical conditions limiting ability to participate in either the Tai Chi or stretching programs as determined by primary care physicians
* Any intra-articular steroid injections in the previous 3 months or reconstructive surgery on the affected knee
* Any intra-articular Synvisc or Hyalgan injections in the previous 6 months
* Inability to pass the Mini-Mental Status examination (with a score below 24)
* Enrollment in any other clinical trial within the last 30 days
* Plan to permanently relocate from the region during the trial period
* Non English Speaking

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Division of Rheumatology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wang C, Collet JP, Lau J. The effect of Tai Chi on health outcomes in patients with chronic conditions: a systematic review. Arch Intern Med. 2004 Mar 8;164(5):493-501. doi: 10.1001/archinte.164.5.493. PMID 15006825
- [Background] Wang C, Roubenoff R, Lau J, Kalish R, Schmid CH, Tighiouart H, Rones R, Hibberd PL. Effect of Tai Chi in adults with rheumatoid arthritis. Rheumatology (Oxford). 2005 May;44(5):685-7. doi: 10.1093/rheumatology/keh572. Epub 2005 Mar 1. No abstract available. PMID 15741197
- [Derived] Wang C, Schmid CH, Hibberd PL, Kalish R, Roubenoff R, Rones R, McAlindon T. Tai Chi is effective in treating knee osteoarthritis: a randomized controlled trial. Arthritis Rheum. 2009 Nov 15;61(11):1545-53. doi: 10.1002/art.24832. PMID 19877092
- [Derived] Wang C, Schmid CH, Hibberd PL, Kalish R, Roubenoff R, Rones R, Okparavero A, McAlindon T. Tai Chi for treating knee osteoarthritis: designing a long-term follow up randomized controlled trial. BMC Musculoskelet Disord. 2008 Jul 29;9:108. doi: 10.1186/1471-2474-9-108. PMID 18664276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the 5-month recruitment period, we screened 366 patients from the Greater Boston area using telephone interviews. 62 potential patients visited the Clinical and Translational Research Center at Tufts Medical Center for further eligibility screening; 40 were eligible after baseline evaluation and randomized to Tai Chi or attention control.
Pre-assignment Details: We excluded individuals with: prior Tai Chi training or similar alternative medicine types like Qi Gong or yoga; serious medical conditions; intra-articular steroid injections in the last 3 months, reconstructive surgery on the affected knee, and intra-articular hyaluronate injections in the previous 6 months; failed the Mini-Mental examination.
Groups:
- Tai Chi: 20 participants were randomly assigned to practice a Tai Chi program based on the classical Yang Style for 60 minutes, twice a week, over 12 weeks.
- Attention Control: 20 participants were randomly assigned to a wellness education and stretching program for the control group, which provided an active control for the attention being paid to the Tai Chi group.
Period: Overall Study
Arm/Group | Tai Chi | Attention Control
Started | 20 | 20
Completed | 20 (No patient withdrew from the study (20/20 participants completed follow-ups at 12, 24 and 48 weeks).) | 20 (No patient withdrew from the study (20/20 participants completed follow-ups at 12, 24 and 48 weeks).)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi | Attention Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.1) | 68 (7.0) | 65 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in the Western Ontario and McMaster University Index (WOMAC) Pain Subscale Between Baseline and 12 Weeks
Description: WOMAC scale range: 0 millimeters (no pain) to 500 millimeters (severe pain), ordinal. Change: score at 12 weeks minus score at baseline. Negative numbers reported here indicate improvement in condition from baseline. (So -100 indicates a 100-point improvement from baseline.)
Time Frame: between baseline and 12 weeks.
Population: We analyzed the data on an intent-to-treat basis.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
mm | -157.25 [-203.11 to -111.39] | -38.45 [-84.31 to 7.41]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = -118.80, 95% CI 2-sided [-183.66 to -53.94]

2. Secondary Outcome: Change in WOMAC Function From Baseline to 12, 24, and 48 Weeks.
Description: The WOMAC is a validated, self-administered instrument specifically designed to evaluate knee and hip OA. The function subscale had a score range 0-1700mm, with higher scores indicating more severe disease. Negative numbers reported here (change in subscale score) indicate improvement in condition from baseline. (So -200 indicates a 200-point improvement from baseline.)
Time Frame: from baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
mm
  12 Week | -506.75 [-640.66 to -372.84] | -182.15 [-316.06 to -48.24]
  24 Week | -440.50 [-574.41 to -306.59] | -257.30 [-391.21 to -123.39]
  48 Week | -405.85 [-539.76 to -271.94] | -300.55 [-434.46 to -166.64]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -324.60, 95% CI 2-sided [-513.98 to -135.22]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -183.20, 95% CI 2-sided [-372.58 to 6.18]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 week; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis; Mean Difference (Final Values) = -105.30, 95% CI 2-sided [-294.68 to 84.08]

3. Secondary Outcome: Change in WOMAC Stiffness From Baseline to 12, 24, and 48 Weeks.
Description: The WOMAC is a validated, self-administered instrument specifically designed to evaluate knee and hip OA. The stiffness subscale has a score range 0-200mm, with higher scores indicating more severe disease. Negative numbers reported here (change in subscale score) indicate improvement in condition from baseline. (So -100 indicates a 100-point improvement from baseline.)
Time Frame: baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
mm
  12 Week | -73.05 [-94.36 to -51.74] | -50.15 [-71.46 to -28.84]
  24 Week | -65.00 [-86.31 to -43.69] | -50.20 [-71.51 to -28.89]
  48 Week | -64.15 [-85.46 to -42.84] | -60.50 [-81.81 to -39.19]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 week; Test type: Superiority or Other; p = 0.1, Mixed Models Analysis; Mean Difference (Final Values) = -22.90, 95% CI 2-sided [-53.04 to 7.24]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 week; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis; Mean Difference (Final Values) = -14.80, 95% CI 2-sided [-44.94 to 15.34]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Week; Test type: Superiority or Other; p = 0.8, Mixed Models Analysis; Mean Difference (Final Values) = -3.65, 95% CI 2-sided [-33.79 to 26.49]

4. Secondary Outcome: Change in WOMAC Pain Scores From Baseline to 24 and 48 Weeks.
Description: The WOMAC is a validated, self-administered instrument specifically designed to evaluate knee and hip OA. The WOMAC was administered to the participants at baseline, 12, 24 and 48 weeks. The pain subscale score range was 0-500mm, with higher scores indicating more severe disease. Negative numbers reported here (change in subscale score) indicate improvement in condition from baseline. (So -200 indicates a 200-point improvement from baseline.)
Time Frame: baseline to 24, 48 weeks
Population: The 12-Week WOMAC scores are listed under Primary Outcome. The 24-Week and 48-Week scores are listed as Secondary Outcomes.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
mm
  24 Weeks | -131.55 [-177.41 to -85.69] | -64.60 [-110.46 to -18.74]
  48 Weeks | -115.35 [-161.21 to -69.49] | -69.20 [-115.06 to -23.34]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -66.95, 95% CI 2-sided [-131.81 to -2.09]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 48 Week; Test type: Superiority or Other; p = 0.2, Mixed Models Analysis; Mean Difference (Final Values) = -46.15, 95% CI 2-sided [-111.01 to 18.71]

5. Secondary Outcome: Change in Patient Global Knee Pain Assessment Visual Analogue Scale (VAS)
Description: Participants completed a self-reported knee-specific global pain VAS with scores ranging from 0 to 10 centimeters (cm); 0 equals no pain. Negative numbers reported here indicate improvement in condition from baseline. (So -10 indicates a 10-point improvement from baseline.)
Time Frame: baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
cm
  12 Week | -2.98 [-4.16 to -1.80] | -0.83 [-2.00 to 0.35]
  24 Week | -2.36 [-3.53 to -1.18] | -1.71 [-2.89 to -0.53]
  48 Week | -1.65 [-2.83 to -0.48] | -1.70 [-2.87 to -0.52]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-3.82 to -0.49]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.4, Mixed Models Analysis; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-2.31 to 1.02]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 weeks; Test type: Superiority or Other; p = 1.0, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.62 to 1.70]

6. Secondary Outcome: Change in Physician Global Knee Pain Assessment Visual Analogue Scale (VAS)From Baseline to 12, 24, and 48 Weeks.
Description: The study physician who was blinded to group assignment completed a global knee pain assessment VAS with scores ranging from 0 to 10cm; 0 equals no pain. Negative numbers reported here indicate improvement in condition from baseline. (So -10 indicates a 10-point improvement from baseline.)
Time Frame: baseline to 12, 24, 48 weeks
Population: Note: Data for only 19 participants in the Attention Control group was analyzed at 48 Weeks due to lack of available data.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
cm
  12 Week | -3.14 [-3.88 to -2.41] | -1.44 [-2.18 to -0.70]
  24 Week | -2.59 [-3.33 to -1.86] | -2.06 [-2.80 to -1.32]
  48 Week | -2.53 [-3.27 to -1.80] | -1.50 [-2.25 to -0.75]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.75 to -0.66]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.58 to 0.51]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Week; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-2.09 to 0.02]

7. Secondary Outcome: Change in Timed Chair Stand From Baseline to 12, 24, and 48 Weeks.
Description: Timed stand tests measure the time taken to complete ten full stands from a sitting position. Patients began the chair stand seated with their arms folded across their chests, then rose to a standing position and sat back down with their back against the back rest of the chair. The test was completed when the patient stood for the tenth repetition. Chair stand time was measured in seconds, with lower scores indicating improved state. Negative numbers reported here indicate improvement in condition from baseline. (So -10 indicates a 10-second improvement from baseline.)
Time Frame: baseline to 12, 24, 48 weeks
Population: Note: Data for only 18 participants in the Attention Control group was analyzed for the 48-week timepoint to do availability of data.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 19 | 19
seconds
  12 Week | -12.03 [-15.60 to -8.46] | -1.15 [-4.70 to 2.40]
  24 Week | -9.87 [-13.44 to -6.30] | -4.75 [-8.30 to -1.20]
  48 Week | -9.22 [-12.79 to -5.65] | -3.24 [-6.85 to 0.37]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.00005, Mixed Models Analysis; Mean Difference (Final Values) = -10.88, 95% CI 2-sided [-15.91 to -5.84]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -5.12, 95% CI 2-sided [-10.15 to -0.08]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Week; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = -5.98, 95% CI 2-sided [-11.06 to -0.91]

8. Secondary Outcome: Change in 6 Minute Walk Test From Baseline to 12, 24, and 48 Weeks.
Description: The 6 minute walk test is a reliable measure of functional exercise capacity. Patients were asked to walk as fast and as far as possible within the 6-minute period and were accompanied by the research staff using a wheel measure that measured distance covered in inches and convereted to yards; higher scores indicated improved state. Higher numbers reported here indicate more improvement from baseline.
Time Frame: baseline to 12, 24, 48 weeks
Population: Note: Data for only 18 patients from Tai chi group was analyzed for 12 week timepoint. Data for 19 patients from the Attention Control group was analyzed at 48 week timepoint.
Measure: Mean (95% Confidence Interval); unit: yards
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 19 | 20
yards
  12 Week | 48.33 [11.15 to 85.50] | -1.76 [-50.70 to 47.18]
  24 Week | 53.12 [10.04 to 96.21] | 9.41 [-33.48 to 52.30]
  48 Week | 35.17 [-17.29 to 87.64] | 20.56 [-20.73 to 61.85]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.1, Mixed Models Analysis; Mean Difference (Final Values) = 50.08, 95% CI 2-sided [-10.34 to 110.50]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Week; Test type: Superiority or Other; p = 0.1, Mixed Models Analysis; Mean Difference (Final Values) = 43.71, 95% CI 2-sided [-15.07 to 102.50]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Weeks; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis; Mean Difference (Final Values) = 14.61, 95% CI 2-sided [-49.36 to 78.59]

9. Secondary Outcome: Change in Standing Balance From Baseline to 12, 24, and 48 Weeks.
Description: The standing balance test included tandem, semi-tandem, side-by-side, and one-legged stands. Patients were asked to maintain each position for 30 seconds. For each task, the research staff first demonstrated the task, asked the patient if they felt comfortable and ready and then supported the patient while positioning themselves. One point was given if they exceeded 30 seconds and none if they could not or did not attempt the test. Higher numbers reported here indicate more improvement from baseline.
Time Frame: baseline to 12, 24, 48 weeks
Population: Note: Data for only 19 patients in Attention Control group was analyzed for 48-week timepoint due to availability of data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
units on a scale
  12 Weeks | 0.15 [-0.16 to 0.46] | 0.25 [-0.06 to 0.56]
  24 Weeks | 0.15 [-0.16 to 0.46] | 0.08 [-0.24 to 0.39]
  48 Weeks | 0.35 [0.04 to 0.66] | 0.46 [0.14 to 0.77]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Weeks; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.54 to 0.34]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Weeks; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.37 to 0.52]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 weeks; Test type: Superiority or Other; p = 0.6, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.55 to 0.34]

10. Secondary Outcome: Change in Center for Epidemiology Studies Depression Index (CES-D)From Baseline to 12, 24, and 48 Weeks.
Description: The CES-D was used to assess depressive symptoms. It included a 20-item Likert-type scale with scores ranging from 0 to 60. Higher scores indicated greater dysphoria. Negative numbers reported here indicate improvement in condition from baseline. (So -1 indicates a 1-point improvement from baseline.)
Time Frame: baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
units on a scale
  12 Week | -7.40 [-10.88 to -3.92] | -0.70 [-4.18 to 2.78]
  24 Week | -6.40 [-9.88 to -2.92] | -1.10 [-4.58 to 2.38]
  48 Week | -7.25 [-10.73 to -3.77] | 1.65 [-1.83 to 5.13]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Week; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = -6.70, 95% CI 2-sided [-11.63 to -1.77]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Weeks; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = -5.30, 95% CI 2-sided [-10.23 to -0.37]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Week; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = -8.90, 95% CI 2-sided [-13.83 to -3.97]

11. Secondary Outcome: Change in Self-Efficacy Scale From Baseline to 12, 24, and 48 Weeks.
Description: Self-efficacy is important for individuals to adopt and maintain a program of regular physical activity. The patient rates his/her confidence of being physically active in different types of situations on a 5-item scale with responses ranging from "not at all confident" to "extremely confident". The total score is coputed by calculating the average of all 5 questions. A higher score indicates greater self-efficacy. Higher numbers reported here indicate more improvement from baseline.
Time Frame: baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
units on a scale
  12 Week | 0.60 [0.12 to 1.08] | -0.11 [-0.59 to 0.37]
  24 Week | 0.68 [0.20 to 1.16] | -0.17 [-0.65 to 0.31]
  48 Week | 0.72 [0.24 to 1.20] | -0.24 [-0.72 to 0.24]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Weeks; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [0.03 to 1.39]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Weeks; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.17 to 1.53]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Weeks; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.28 to 1.64]

12. Secondary Outcome: Change in Medical Outcome Study Short Form 36 (SF-36) Physical Component From Baseline to 12, 24, and 48 Weeks.
Description: Health related quality of life assessments were made using the SF-36. The SF-36 measures 8 domains: physical functioning, role-physician, bodily pain, general health, vitality, social function, emotional health and mental health. The Physical Component of the SF-36 had scores that ranged from 0 to 100; 0 equals worst health state. Change: Higher numbers reported here indicate more improvement in condition from baseline.
Time Frame: baseline, 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
units on a scale
  12 Weeks | 11.57 [8.08 to 15.06] | 4.14 [0.65 to 7.63]
  24 Weeks | 10.80 [7.31 to 14.29] | 6.29 [2.80 to 9.77]
  48 Weeks | 10.41 [6.92 to 13.90] | 4.10 [0.61 to 7.58]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Weeks; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 7.43, 95% CI 2-sided [2.50 to 12.36]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Weeks; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = 4.51, 95% CI 2-sided [-0.42 to 9.45]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Weeks; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 6.32, 95% CI 2-sided [1.38 to 11.25]

13. Secondary Outcome: Change in Medical Outcome Study Short Form 36 (SF-36) Mental Component
Description: Health related quality of life assessments were made using the SF-36. The SF-36 measures 8 domains: physical functioning, role-physician, bodily pain, general health, vitality, social function, emotional health and mental health. The Mental Component of the SF-36 had scores that ranged from 0 to 100; 0 equals worst health state. Change: Higher numbers reported here indicate more improvement in condition from baseline.
Time Frame: baseline to 12, 24, 48 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Attention Control
Number analyzed (Participants) | 20 | 20
units on a scale
  12 Weeks | 2.14 [-2.35 to 6.64] | 1.93 [-2.56 to 6.43]
  24 Weeks | 4.39 [-0.11 to 8.89] | 4.50 [0.00 to 9.00]
  48 Weeks | 5.80 [1.31 to 10.30] | 1.04 [-3.46 to 5.53]
Statistical Analysis 1: Comparison: Tai Chi vs Attention Control; 12 Weeks; Test type: Superiority or Other; p = 0.9, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-6.15 to 6.57]
Statistical Analysis 2: Comparison: Tai Chi vs Attention Control; 24 Weeks; Test type: Superiority or Other; p = 1.0, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-6.47 to 6.25]
Statistical Analysis 3: Comparison: Tai Chi vs Attention Control; 48 Weeks; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis; Mean Difference (Final Values) = 4.77, 95% CI 2-sided [-1.59 to 11.13]

ADVERSE EVENTS:
Time Frame: during 12 week intervention period
Description: One participant in the Tai Chi group reported an increase in knee pain at the 2 week assessment. This was resolved following modification of that participant's Tai Chi technique.
Arm/Group | Tai Chi | Attention Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi (N=20) | Attention Control (N=20)
increased knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant in the Tai Chi group reported an increase in knee pain at the 2 week assessment. This was resolved following modification of that participant's Tai Chi technique.

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The contents of this manuscript are solely the responsibility of the authors and do not necessarily represent the official views of the National Center for Complementary and Alternative Medicine or the National Institutes of Health. The sponsors had no role in the design and conduct of the study; collection, management, analysis, and interpretation of the data; and preparation, review or approval of the manuscript.